CLINICAL TRIAL: NCT04486560
Title: Safety of a Sheath Cryoprobe Bronchoscopic Transbronchial Biopsy Technique (The FROSTBITE Trial)
Brief Title: Safety of a Sheath Cryoprobe Bronchoscopic Transbronchial Biopsy Technique
Acronym: FROSTBITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00235679
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Lung Diseases
Keywords: lung; cryoprobe; bronchoscopic; biopsy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: This is a multi-center, non-randomized, single-arm, prospective trial. Therefore, all participants will have their transbronchial biopsy with the 1.1mm sheath cryoprobe rather than forceps or another currently available larger cryoprobe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm: Cryoprobe (Experimental): Everyone who enrolls in this study will undergo a standard of care bronchoscopy with a transbronchial biopsy using the 1.1mm sheath cryoprobe.
  Interventions: Device: ERBECRYO® 2 Cryosurgical Unit and Accessories - K190651

INTERVENTIONS:
Device: ERBECRYO® 2 Cryosurgical Unit and Accessories - K190651 — ERBE 1.1mm flexible single-use cryoprobe with oversheath

SUMMARY:
The purpose of this study is to evaluate the safety and collect data on the initial effectiveness of a 1.1mm flexible single-use cryoprobe with oversheath used for transbronchial lung biopsy via a bronchoscopic approach.

DETAILED DESCRIPTION:
A smaller (1.1mm), flexible, single-use cryoprobe with an oversheath has been developed that can be used for transbronchial biopsies. This device has the potential to gather larger and higher quality tissue samples than the standard method using forceps, and with potentially fewer complications than older, larger versions of the cryoprobe.

This study does not involve randomization or assigning different patients to different procedures to compare. Everyone who enrolls in this study will undergo a standard of care bronchoscopy with a transbronchial biopsy using the 1.1mm sheath cryoprobe. The only difference from the standard of care approach is that the physician performing the transbronchial biopsy will use the 1.1mm sheath cryoprobe rather than forceps or another currently available larger cryoprobe.

Patients enrolled in this study will have data collected by research staff for up to 30 days after the bronchoscopic biopsy procedure is performed. This 30-day follow-up period is the standard of care following bronchoscopic biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, ≥ 18-years-old
* Scheduled to undergo bronchoscopy with transbronchial biopsy as the standard medical care determined by their treating pulmonologist

Exclusion Criteria:

* Pregnant or nursing females, or females of child bearing potential who refuse to take a pregnancy test prior to enrollment
* Individuals with current or recent systematic conditions, such as uncontrolled hypertension (systolic > 200 mmHg or diastolic > 110 mmHg), type 1 diabetes, severe pulmonary hypertension, acute kidney injury, stroke (within the last 6 months) or myocardial infarction (within the last 3 months)
* Presence of bleeding disorder
* Platelet count <50,000
* Current use of systemic anticoagulation or antiplatelet therapy without the ability to hold therapy for the recommended amount of time prior to an invasive procedure (aspirin monotherapy is acceptable)
* International Normalized Ratio (INR) <1.5
* Robotic Bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm: Cryoprobe
Started | 51
Completed | 50
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26 (7)
Smoking Status [Count of Participants; unit: Participants]
  Never | 28
  Current | 2
  Former | 20
Indication for Biopsy [Count of Participants; unit: Participants]
  Pulmonary Parenchymal Lesion | 3
  Diffuse Lung Disease | 22
  Lung Transplant | 25
Type of Airway [Count of Participants; unit: Participants]
  Laryngeal Mask Airway | 19
  Endotracheal Tube | 21
  Rigid Bronchoscopy | 10
Bronchial Blocker Used [Count of Participants; unit: Participants] — Participants in whom bronchial blocker was used.
  Participants | 8
Location of Biopsy [Count of Participants; unit: Participants]
  Right Upper Lobe | 2
  Right Middle Lobe | 2
  Right Lower Lobe | 31
  Left Upper Lobe | 3
  Left Lower Lobe | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: The number of participants enrolled who experienced a device related Serious Adverse Events (SAEs). SAEs include Grade 3-4 bleeding (bleeding causing cardiopulmonary instability or requiring inflation of a bronchial blocker), pneumothorax requiring chest tube placement (Grade 2+), or 30-day respiratory failure and death.
Time Frame: Within 30 days of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: Number of Participants With Minor Adverse Events
Description: The number of participants enrolled who experienced a device related Minor Adverse Event (AE). AEs include Grade 1-2 bleeding (bleeding requiring suction to clear or wedging of the biopsied segment with the flexible bronchoscope and/or iced saline), or pneumothorax not requiring chest tube placement (Grade 1).
Time Frame: Within 30 days of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Participants
  Grade 1 Pneumothorax | 2
  Grade 1-2 Bleeding | 25

3. Secondary Outcome: Mean Histologic Accessibility Grade
Description: Grade 0: Does not contain alveolar structures and can therefore not be assessed
  Grade 1: Very poor specimen quality; not possible to assess the relevant morphologic and histologic features
  Grade 2: Poor specimen quality; assessment of relevant morphologic and histologic structures and features is severely compromised and not possible
  Grade 3: High limitations in specimen quality; assessment is severely compromised but limited evaluation is possible
  Grade 4: Moderate limitations in specimen quality; assessment is moderately compromised but evaluation is possible
  Grade 5: Low limitations in specimen quality; assessment is somewhat compromised but possible
  Grade 6: The specimen allows for complete and unrestricted assessment of all relevant morphologic and histologic structures and features
Time Frame: Data assessed at the time of review of biopsy sample (up to one year post index procedure) and participants were assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
score on a scale | 4.9 (1.3)

4. Secondary Outcome: Diagnostic Yield as Assessed by Number of Patients for Which Cryobiopsy Led to a Diagnosis
Description: Diagnostic yield is defined as number of patients for which cryobiopsy led to a diagnosis. Diagnostic yield will be determined from the results of cryobiopsy specimen only. A biopsy that results in a specific diagnosis, either malignant or benign (granuloma, inflammation, fibrosis, infection) will be assumed to be a true positive. Atypia, minimal inflammation or lung parenchyma without pathologic findings on final pathology reads are considered non-diagnostic.
Time Frame: During procedure, up to 1 hour
Population: The analysis was broken down by type of cryobiopsy indication.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Participants
  Lung Transplant: number analyzed (Participants) | 25
  Lung Transplant | 23
  Diffuse Lung Disease: number analyzed (Participants) | 22
  Diffuse Lung Disease | 16
  Pulmonary Parenchymal Lesion: number analyzed (Participants) | 3
  Pulmonary Parenchymal Lesion | 1

5. Secondary Outcome: Total Histologic Area (Square Millimeters)
Description: Amount of total histologic tissue in square millimeters observed under microscope.
Time Frame: as for outcome 3
Measure: Mean (Full Range); unit: square millimeters
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
square millimeters | 54.4 [21.1 to 87.7]

6. Secondary Outcome: Alveolated Area (Square Millimeters)
Description: Total amount of area in square millimeters containing alveoli.
Time Frame: as for outcome 3
Measure: Mean (Full Range); unit: square millimeters
Units Other Than Participants: Number of Pieces
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Number analyzed (Number of Pieces) | 231
square millimeters
  Per Patient | 11.39 [0 to 51.6]
  Per Piece | 2.47 [0 to 18.47]

7. Secondary Outcome: Open Alveoli Percent
Description: Percentage of all alveoli that are open.
Time Frame: as for outcome 3
Measure: Mean (Full Range); unit: percent
Units Other Than Participants: Number of Samples
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Number analyzed (Number of Samples) | 182
percent | 66.48 [0 to 100]

8. Secondary Outcome: Percent Crush Artifact
Description: Percent of tissue distortion resulting from even the minimal compression of the tissue, which may rearrange tissue morphology.
Time Frame: as for outcome 3
Measure: Mean (Full Range); unit: percent
Units Other Than Participants: Number of samples
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Number analyzed (Number of samples) | 190
percent | 0.5 [0 to 90]

9. Secondary Outcome: Artifact Free Lung Parenchyma Percent
Description: Percent of the lung parenchyma (alveoli, alveolar ducts and respiratory bronchioles) without artifact.
Time Frame: as for outcome 3
Measure: Mean (Full Range); unit: percent
Units Other Than Participants: Number of Samples
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
Number analyzed (Number of Samples) | 181
percent | 90.86 [0 to 100]

10. Secondary Outcome: Activation Time (Seconds)
Description: Time of activation of cryoprobe.
Time Frame: At the time of procedure, up to 1 hour
Measure: Mean (Full Range); unit: seconds
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
seconds | 4.2 [3.2 to 5.2]

11. Secondary Outcome: Procedure Time
Description: Time for entire procedure measured in minutes.
Time Frame: At the time of procedure, up to 1 hour
Measure: Mean (Full Range); unit: minutes
Arm/Group | Single Arm: Cryoprobe
Number analyzed (Participants) | 50
minutes | 22 [10 to 38]

ADVERSE EVENTS:
Time Frame: Day of procedure through 30 days post-procedure
Description: Primary Safety Endpoint Serious Adverse Event: Occurrence of bleeding grade ≥ 3, pneumothorax grade ≥ 2, post-procedure respiratory failure, and/or death related to the device.
  Secondary Safety Endpoint Serious Adverse Event: Occurrence of bleeding grade < 3 and/or pneumothorax grade < 2 related to the device.
Arm/Group | Single Arm: Cryoprobe
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 22/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Cryoprobe (N=50)
SECONDARY SAFETY ENDPOINT Adverse Event (Respiratory, thoracic and mediastinal disorders) | 22 (22) — Occurrence of bleeding grade < 3 and/or pneumothorax grade < 2 related to the device

LIMITATIONS AND CAVEATS:
All procedures were performed at large academic centers so procedural volume and pathology may not be generalizable. Larger proportion of lung transplant patients enrolled means there is a lack of heterogeneity in disease entities. Study aimed to address safety so the design and sample size is too small to accurately estimate diagnostic yield. Sheath was required for all cases, precluding use of robotic-assisted bronchoscopy (and underrepresentation of lung cancer).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04486560/Prot_SAP_000.pdf